CLINICAL TRIAL: NCT03171324
Title: a Randomized Control Trial to Assess the Effect of Early vs Routine Iron Supplementation on Iron Store and Growth in Term Small for Gestational Age and Appropriate for Gestational Age Infants at 1 Year
Brief Title: to Assess the Effect of Early vs Routine Iron Supplementation on Iron Store and Growth in Term Infants
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Deepanjan Bhattacharya (Other)
Collaborators: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Sponsor-Investigator, Deepanjan Bhattacharya, PRINCIPAL INVESTIGATOR Junior resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Deep1234
Record Dates: First submitted 2017-02-26; First posted 2017-05-31 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Iron-Dextran Complex

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- AGA 6 weeks (Experimental): Iron supplementation will be started at 2mg/kg from 6 weeks of age to 1 year
  Interventions: Drug: Iron Supplement
- AGA 6 months (Experimental): Iron supplementation will be started from 6 months of age to 1 year
  Interventions: Drug: Iron Supplement
- SGA 6 weeks (Experimental): Iron supplementation will be started from 6 weeks of age to 1 year
  Interventions: Drug: Iron Supplement
- SGA 6 months (Experimental): Iron supplementation will be started from 6 months of age to 1 year
  Interventions: Drug: Iron Supplement

INTERVENTIONS:
Drug: Iron Supplement — 2 mg/kg/day elemental iron
  Other Names: Tonoferon

SUMMARY:
Term infants (Small for Gestational Age and Appropriate for Gestational Age) would be randomized to receive oral iron supplementation from 6 weeks and 6 months. Growth in terms of Occipitofrontal circumference, length and weight would be monitored at 6 weeks, 6 months and 1 year of age. Hemoglobin, RBC (Red blood corpuscles) indices and ferritin would be monitored at 6 months and 1 year of age.

DETAILED DESCRIPTION:
Study Design: Randomized Controlled Trial, Open label. Study setting: Neonatology unit, Postnatal clinic and children Out Patient Department and growth clinic at Advanced Pediatrics Centre, Postgraduate Institute of Medical Education and Research (PGIMER) Chandigarh Study period: January 2017 to June 2018 Consecutively born all term babies in the labour room, PGIMER,Chandigarh, and residing in tricity area and within 100 km radius of Chandigarh will be screened for fulfilment of inclusion criteria within 1st 24 hours of life. Babies will be classified as SGA or AGA as per Fenton's growth chart.

Details of maternal and neonatal characteristics will be recorded in a structured proforma with a verbal consent of parents and counselling for follow up from 6 weeks onwards till 1 year of age. Details of discharge characteristics and anthropometry will be recorded in a structured format. Exclusive breast feeding till 6 months will be advised to all mothers. Kuppuswamy's scale will be used to assess socioeconomic status.

Birth details of babies will be recorded from the labour room register in PGIMER Labour Room. Their parents will be asked to report to the PostNatal Clinic after 6 weeks for their routine followup. Inclusion and exclusion criteria will be applied at the postnatal visit at 6 weeks, and consent will be taken. Randomisation will be done at 6 weeks in the postnatal clinic, along initiation of iron in the early (6 weeks group) These babies are routinely followed up in Post Natal Clinic (PNC) at 6 weeks for maternal check up and for initiation of vaccination. Subsequently they are seen in Children's OPD at 10 and 14 wks to complete vaccination and at 6 months for complementary feeding advice.

A written, informed consent would be obtained from one of the parents after explaining details of intervention at enrolment at 6 weeks.

Currenly as per unit protocol, all term babies receive only Vitamin D drops 400 IU daily for 1 year. No other supplements are given till 6 months.

Infants in early group will receive iron supplementation from 6 weeks of age, while those in routine group will receive iron supplementation from 6 months of age as per World Health Organisation (WHO) guidelines.

This will be an open label study regarding group allocation due to nature of the study however labs will be blinded.

Ethics permission will be sought from Institute Research ethics committee as per protocol.

RANDOMIZATION Term SGA and AGA babies fulfilling the inclusion criteria would be randomised to early and routine iron supplementation using computer generated random numbers using block randomization in opaque sealed envelopes which will be opened once the parental consent is given. Flow of patients will be recorded as per CONSORT guidelines.

Randomization will be done in 2 separate groups (AGA and SGA).

Patients along with their parents would be contacted on phone at 6 weeks to report to PNC along with their mothers where enrolment and randomization will take place. Subsequently babies will be seen at 10 weeks, 14 weeks, 6 months , 9 months and 1 yr of age . Compliance would be ensured by telephonic conversation in the interim period. Parents will be taught to use daily alarms in mobile for administration of iron.

At each visit they will be examined by PI and the supervising consultant in CHOPD for Anthropometry, Feeding/ Diet, Any illness, Compliance about drug intake and Drug dose adjustments.

At 6 months, parents would be advised to give complementary feeding as per CF chart.

Iron supplementation would be started at 3 mg/kg/day at 6 weeks in early group as well as 6 months group using a liquid preparation of iron, vitamin B12 and folic acid.

Composition per 1 ml Elemental iron 25 mg + lysine hydrochloride 200 mg + Vitamin B12 5 mcg + Folic acid 200 mcg

If the child suffers from any illness during study period, it shall be noted. Sampling for ferritin will not be done at time of illness; it will be done 1 week after illness.

Any additional drug intake by the child during this period will also be noted in the proforma.

All illnesses including all OPD visits and admissions during study period will be recorded.

Details of complementary feeding would be taken by 24 hour recall method, and calculation of calorie and protein intake per day would be done.

HEMATOLOGICAL PARAMETERS Blood samples would be drawn at 6 months of age in all babies and repeated at 1 year of age. 2 ml of blood would be drawn by aseptic precautions in 1 EDTA vial for Hemoglobin, RBC indices as well as ferritin.. No payment will be required to be made, as it will be purchased from departmental research grant.

The collected EDTA sample would be first processed for hemogram by 6-part differential Sysmex XN-1000 (Japan) automatic analyser which would use 400 microlitre of blood. Processing would be done on a daily basis. Reports will be collected by the primary investigator in the evening and will be handed over to the parents during followup.

The EDTA sample would then be centrifuged at 300 rpm for 10 minutes to separate the plasma, which will be kept in properly labelled 2ml Eppendorf tubes. The samples would be stored at -20°C at APC 4A Hematology Lab. Processing would be done in batches every 2nd day by chemiluminescence assay using ADIVA Centaur Ferritin assay.

Samples for hemogram and ferritin will be processed under the guidance of coguide Dr. Prateek Bhatia.

GROWTH ASSESSMENT Growth assessment would be done by the principal investigator under the guidance of Prof AK Bhalla at 6 weeks, 6 months and 1 year of age, in Growth Lab, APC 5D.

1. WEIGHT: The nude body weight of each child in standing /lying down position will be recorded on an electronic weighing scale (make Every India Limited) upto accuracy of 50 gram. Scale is calibrated before each individual weighing then weight will be plotted on WHO growth charts [ANNEXURE 8], and the respective percentile noted
2. LENGTH: Infantometer will be used to measure crown heel length up to an accuracy of 1 mm. Each infant will be placed over the horizontal board. The infant's head will be adjusted against the head plate so that the lower orbital margin and tragus lie on the same plane. The knee of the infant will be straightened and the foot will push the foot plate out so that the there is no gap between the foot and the foot plate. The reading in the tape across at the level of the foot plate will be noted after taking the infant out. Length will be plotted on WHO growth chart [ANNEXURE 9], and the respective percentile noted.
3. HEAD CIRCUMFERENCE: Head circumference (HC) will be measured by using non flexible fibre glass tape with minimum record of 1mm. The measure will be taken by encircling the tape firmly around the head just above the supra orbital ridges and over the most prominent backwardly protruding part of the occiput. HC will be plotted on WHO growth chart [ANNEXURE 10], and the respective percentile noted.

Standard deviation scores for weight, length and HC scores for corrected age will be calculated using the WHO anthro for PC software.

Children will be assessed at

* 6 weeks - anthropometry (length, weight, HC) at enrolment and randomization
* 6 months - anthropometry and haematological parameters (Hemoglobin, RBC indices, Ferritin)
* 1 year - anthropometry and haematological parameters (Hemoglobin, RBC indices, Ferritin)

STUDY ENDPOINTS

1. At 1 year
2. Any condition requiring blood transfusion before 1 year

PRIMARY OUTCOME - 1. Proportion of infants with Iron Deficiency Anemia. at 6 months and 1 year in 2 groups

SECONDARY OUTCOME -

1. Growth parameters ( weight, length and HC and their z scores) in 2 groups at 6 months and 1 year Serum ferritin in early vs routine iron supplementation group at 6 months and 1 year All the above outcomes will be assessed in SGA and AGA groups separately.

IRON DEFICIENCY will be defined as serum ferritin < 15 µg/l. IRON DEFICIENCY ANEMIA will be defined as Iron deficiency (serum ferritin < 15 µg/l) with haemoglobin less than the age specific cutoffs.

ELIGIBILITY:
Inclusion Criteria:

* Term infants (born after 37 completed weeks of gestation by USG dating or LMP and postnatally by New ballard scoring whichever applicable)
* Appropriate for gestational age (as per revised Fenton's chart 2013)
* Small for gestational age (birth weight <10th percentile as per revised Fenton's chart 2013) - Parents consenting to follow up till 1 year
* Parents residing within 100 kilometres of Chandigarh

Exclusion Criteria:

1. H/o blood product transfusion prior to study enrolment
2. Neonatal jaundice due to hemolytic anemia
3. Severe birth asphyxia defined as 1 minute Apgar score 0-3 with or without moderate to severe HIE (Hypoxic Ischemic Encephalopathy).
4. Severe sepsis with septic shock
5. Suspect haematological disorders
6. Infants with chronic diseases like congenital heart disease, cholestatic jaundice and suspected liver disease, suspected or diagnosed renal tubular acidosis, suspected or diagnosed inborn errors of metabolism
7. Suspected or proven chromosomal abnormalities.

Ages: 6 Weeks to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Iron deficiency anemia | 1 year
  Hemoglobin

SECONDARY OUTCOMES:
Growth parameter1 | 6 months
  Occipitofrontal circumference (OFC) in cm at 6 months
Growth parameter2 | 6 months
  Length (in cm) at 6 months
Growth parameter3 | 6 months
  Weight (in kg) at 6 months
Iron stores | 6 months
  iron stores will be evaluated by ferritin, and anemia evaluated by hemoglobin
Growth parameter4 | 1 year
  OccipitoFrontal Circumference (in cm) at 1 year of age.
Growth parameter5 | 1 year
  Length (in cm) at 1 year of age.
Growth parameter6 | 1 year
  Weight (in kg) at 1 year of age.
Iron stores | 1 year
  iron stores will be evaluated by ferritin at 1 year of age, along with hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Kanya Mukhopadhyay, MD DM, Study Director — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No
Not to be shared